CLINICAL TRIAL: NCT03354650
Title: Epidemiology of Neonatal Sepsis in Infants Admitted to Neonatal Intensive Care Unit in Assiut University Children Hospital
Brief Title: Epidemiology of Neonatal Sepsis in Neonatal Intensive Care Unit in Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MSHAhmed, Principal Investigator, Assiut University
Other Study IDs: EONI
Record Dates: First submitted 2017-10-28; First posted 2017-11-28 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Neonatal SEPSIS
MeSH Terms: conditions — Neonatal Sepsis | interventions — Blood Culture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- complete blood count: blood sample is collected from infant to detect presence of sepsis
  Interventions: Diagnostic Test: blood culture
- c reactive protein: measuring c reactive protein in blood sample to determine neonatal sepsis
  Interventions: Diagnostic Test: blood culture

INTERVENTIONS:
Diagnostic Test: blood culture — blood culture to determine causative organisms of neonatal sepsis
  Other Names: other cultures if needed

SUMMARY:
Neonatal sepsis is an important cause of morbidity and mortality in the pediatric age group . It is one of the leading causes of death in the first 28 days of life both in the developed and developing countries.

DETAILED DESCRIPTION:
More than 40% of under-five deaths globally occur in the neonatal period, resulting in 3.1 million newborn death each year.

The majority of these deaths usually occur in low income countries . On the other hand, the survivors of neonatal sepsis are vulnerable to short- and long term neurodevelopmental morbidity .

Neonatal sepsis is a clinical syndrome characterized by signs and symptoms of infection with or without accompanying bacteremia in the first month of life. It includes various systemic infections of the newborn such as septicemia, meningitis, pneumonia, arthritis, osteomyelitis, and urinary tract infections. Superficial infections like conjunctivitis and oral thrush are usually not included under neonatal sepsis.

Diagnosis of sepsis in neonates is challenging due to nonspecific signs and symptoms. The salient clinical features include systemic signs of infection such as fever, hypothermia, tachycardia, failure to thrive, lethargy, irritability, restlessness In addition, laboratory diagnosis until recently was time-consuming. This, therefore, necessitates the initiation of empirical antibiotic therapy pending a definitive diagnosis .

Neonatal sepsis is caused by Gram-positive and Gram-negative bacteria and Candida. The diversity of organisms causing sepsis varies from region to another and changes over time even in the same place .

ELIGIBILITY:
Inclusion Criteria:

• All admitted inborn and out born neonates during this study period will be screened for sepsis

Exclusion Criteria:

• All cases that mimic neonatal sepsis such as;

* Inborn errors of metabolism
* Congestive heart failure
* Hemolytic Disease of Newborn
* Hypoxic ischemic encephalopathy
* Congenital Diaphragmatic Hernia
* Intra cranial hemorrhage
* Respiratory Distress Syndrome

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All admitted male and female infant from the birth to the day 30 after birth
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of neonatal sepsis | up to 4 months
  by measuring the incidence of neonatal sepsis helping to know the size of the problem of neonatal sepsis
prevalence of neonatal sepsis | up to 4 months
  by measuring the prevalence of neonatal sepsis this help us to manage neonatal sepsis accordingly

SECONDARY OUTCOMES:
risk factors and causative organisms of neonatal sepsis | up to 4 months
  by determining the relation between risk factors and incidence of neonatal sepsis and by determining the causative organisms this help in prevention and management of neonatal sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Gehan Mo Kamal El_Din, Professor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided